CLINICAL TRIAL: NCT01884844
Title: Randomized Double-Blind Placebo-Controlled Pilot Study of Vitamin D Supplementation for the Treatment of Bipolar Depression
Brief Title: Vitamin D Supplementation for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Wendy Marsh, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NARSADYI13-15
Record Dates: First submitted 2013-06-17; First posted 2013-06-24 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Bipolar Disorder; Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3, Cholecalciferol, 5000IU po qday for 12 weeks
  Interventions: Drug: Vitamin D3, Cholecalciferol
- Placebo (Placebo Comparator): methylcellulose po qday for 12weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3, Cholecalciferol
  Arms: Vitamin D3
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to whether vitamin d supplementation in those with low levels may reduce depression symptoms in people experiencing bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18years old
* Bipolar disorder (I,II or NOS),
* MADRS Score>7 (mild),
* 25(OH)D level <30ng/ml (insufficient).
* able to take the prescribed vitamin D by mouth

Exclusion Criteria:

Systemic diseases such as:

* liver and kidney diseases,
* known parathyroid disorder,
* disorders of vitamin D metabolism,
* taking vitamin D replacement therapy,
* fat digestion disorder,
* diabetes mellitus,
* gi surgery
* If the serum calcium in the range 2.50-2.55 mmol L, inclusion required a serum PTH below 5.0 pmol L-acute psychiatric urgency:
* active suicidality,
* acute psychosis,
* active substance use<6mo or
* pregnant or nursing females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Marsh, MD MSc, Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - University of Massachusettes, Worcester, Massachusetts
  - University of Massachusetts School of Medicine, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3: Vitamin D3, Cholecalciferol, 5000IU po qday for 12 weeks
  Vitamin D3, Cholecalciferol
- Placebo: methylcellulose po qday for 12weeks
  Placebo
Period: Overall Study
Arm/Group | Vitamin D3 | Placebo
Started | 16 | 17
Completed | 13 | 12
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.3) | 43.3 (12.9) | 44.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 15 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Åsberg Depression Rating Scale
Description: Montgomery-Åsberg Depression Rating Scale Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
  Usual cutoff points are:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: baseline and at 12 week completion
Population: Comparison of bimonthly scale measurements (MADRS, between treatment groups over time were done fitting individual Generalized Linear Models (GLMs) using the initial baseline measurement as an adjustment. Significance was fixed at 0.05%. SPSS v. 23 used
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 12 | 13
units on a scale | 9.4 [3.5 to 15.6] | 6.4 [2.3 to 10.6]
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.89, Fisher Exact

ADVERSE EVENTS:
Time Frame: 12weeks of study
Arm/Group | Vitamin D3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 10/16 | 9/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vitamin D3 (N=16) | Placebo (N=17)
xerostomia (Gastrointestinal disorders) | 4 | 3
appetite decrease (Gastrointestinal disorders) | 3 | 2
diarhea (Gastrointestinal disorders) | 2 | 2
weakness (General disorders) | 3/13 | 3
mild confustion (General disorders) | 2/13 | 2
headache (Nervous system disorders) | 3/13 | 1
mild sedation (General disorders) | 3 | 2
sexual dysfunction, any (Reproductive system and breast disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No